CLINICAL TRIAL: NCT03712423
Title: A Clinical Phase I, Open-label, PET Study With [89Zr]-Df-CriPec® Docetaxel in Patients With Solid Tumours to Assess Biodistribution and Tumour Accumulation of [89Zr]-Df-CriPec® Docetaxel
Brief Title: PET Study With [89Zr]-Df-CriPec® Docetaxel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Cristal Therapeutics (Industry)
Responsible Party: Principal Investigator, C. Menke- van der Houven van Oordt, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-003664-12
Record Dates: First submitted 2017-10-03; First posted 2018-10-19 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Solid Tumor
Keywords: Nanoparticles; Positron-Emission Tomography; Docetaxel; Neoplasms; Quantification
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase I, open-label, single centre immune-PET study with [89Zr]-Df-CriPec® docetaxel in patients with solid tumours to assess biodistribution and tumour accumulation of [89Zr]-Df-CriPec® docetaxel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients [89Zr]-Df-CriPec® docetaxel (Experimental): Day 1 of the Run-in a low dose of [89Zr -Df-CriPec® docetaxel (corresponding to 0.1- 2 mg docetaxel). On Cycle 1 Day 1, the patients will receive unlabelled CriPec® docetaxel of a variable dose up to 60mg/m2 followed < 2 h by a second low dose of [89Zr]-Df-CriPec® docetaxel. On day 1 of each subsequent cycle, patients will only receive unlabelled CriPec® docetaxel . The dose will be the same as was given on Cycle 1 Day 1. For the following patients the dose of unlabelled CriPec® docetaxel combined with the low dose of [89Zr]-Df- CriPec® docetaxel will be variable but never exceed the highest dose of unlabelled CriPec® docetaxel that was determined to be safe in the phase I NAPOLY trial (CT-CL01).
  Interventions: Drug: Cripec Docetaxel

INTERVENTIONS:
Drug: Cripec Docetaxel — 89 Zirconium Cripec Docetaxel PET
  Other Names: 89 Zirconium Cripec Docetaxel PET

SUMMARY:
A clinical phase I, open-label PET study with [89Zr]-Df-CriPec® docetaxel in patients with solid tumours to assess biodistribution and tumour accumulation of [89Zr]-Df-CriPec® docetaxel.

DETAILED DESCRIPTION:
After patient inclusion an fludeoxyglucose-18 ([18F]-FDG) PET scan will be performed to delineate viable tumour lesions. On day 1, patients will receive a low dose of [89Zr]-Df-CriPec® docetaxel (corresponding to approximately 0.1-1 mg docetaxel) followed by maximally 3 [89Zr] PET scans (timing of PET scan can be adapted depending on results obtained, within timeframe of 2 h - 9 days after administration) to evaluate biodistribution and tumour uptake. Two weeks later, the patients will receive unlabelled CriPec® docetaxel up to the Recommended Phase II Dose (RP2D) given every 3 weeks (Q3W) that will be determined in the phase I NAPOLY trial (CT-CL01), immediately followed by a second low dose of [89Zr]-Df-CriPec® docetaxel and maximally 3 [89Zr]PET scans (timing of PET scan can be adapted depending on results obtained, within timeframe of 2 hrs - 9 days after administration) to evaluate biodistribution and tumour uptake with therapeutic dosage.

ELIGIBILITY:
Inclusion Criteria

To be eligible to participate in this study, candidates must meet the following eligibility criteria:

1. Age ≥ 18 years 2 A pathologically confirmed diagnosis of advanced, recurrent and progressive cancer that is refractory to standard therapy or for which no standard therapy exist and where treatment with a taxane is an appropriate treatment option 3. Measurable or evaluable disease according to RECIST criteria v.1.1 Patient must have at least one measurable lesion with a short axis diameter of ≥ 2 cm.

4. Performance status (WHO scale/ ECOG) ≤ 1 (appendix 2) 5. Estimated life expectancy of at least 12 weeks 6. Toxicities incurred as a result of previous anti-cancer therapy (radiation therapy, chemotherapy, or surgery) must be resolved to ≤ grade 2 (as defined by CTCAE version 4.0) 7. ANC ≥ 1.5 x10E9/L; platelets ≥ 100 x 10E9/L; Haemoglobin ≥ 6.0 mmol/L (≥ 9.6 g/dL) 8. Creatinine ≤ 1.5 x upper limit of normal (ULN); or creatinine clearance ≥ 60 mL/ min (Cockcroft-Gault) 9 Serum bilirubin ≤1.5 x ULN, alkaline phosphatase, ASAT and ALAT ≤ 2.5 x ULN, unless related to liver metastases, in which case ≤ 5x ULN is allowed 10 Written informed consent according to local guidelines

Exclusion Criteria

Candidates will be excluded from study entry if any of the following exclusion criteria are met:

1. Less than 4 weeks since the last treatment with other anti-cancer therapies, (i.e. endocrine therapy, immunotherapy, radiotherapy, chemotherapy, etc.), less than 8 weeks for cranial radiotherapy, and less than 6 weeks for nitrosoureas and mitomycin C prior to first study treatment.
2. A history of skin toxicity as a result of prior treatment with taxanes
3. If excessive sequestering of [ 89 Zr] CriPec®docetaxel in healthy liver is observed in the first 3 patients, patients with only liver lesion will not be eligible.
4. Current or recent (within 28 days of first study treatment) treatment with another investigational drug or participation in another investigational study.
5. Active or symptomatic brain metastases. Patients must be on a stable or deceasing dose of corticosteroids and/ or have no requirement for anticonvulsants for 5 days prior to Cycle 1 Day 1.
6. Current malignancies at other sites, with exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin
7. Major surgical procedure (including open biopsy, excluding central line IV and port-a- cath) within 27 days prior to the first study treatment, or anticipation of the need for major surgery during the course of the study treatment
8. Uncontrolled hypertension (systolic >150 mmHg and/ or diastolic > 100 mmHg)
9. Grade ≥ 2 motor or sensory neuropathy symptoms (as defined by CTCAE version 4.03)
10. Known hypersensitivity to any of the study drugs or excipients or taxanes
11. Any active skin condition associated with impaired skin integrity exposing the patient at risk to develop skin toxicity 12 Clinically significant (i.e. active) cardiovascular disease defined as:

    * Stroke within ≤ 6 months prior to first study treatment;
    * Transient Ischemic Attack (TIA) within ≤ 6 months prior to first study treatment ;
    * Myocardial infarction within ≤ 6 months prior to first study treatment;
    * Unstable angina;
    * New Yotk Heart Association (NYHA) Grade II or greater Congestive Heart Failure (CHF);
    * Serious cardiac arrhythmia requiring medication;
    * Clinically relevant pathologic findings in electrocardiogram (ECG)
    * Left ventricle Ejection Fraction (LVEF) by MUGA or ECHO < 50% 13 Patients who are pregnant or breastfeeding 14 Absence of effective means of contraception as of Run-in Day 1 in female patients of childbearing potential (defined as < 2 years after last menstruation and not surgically sterile) ore in male patients who are not surgically sterile and who have female partners if childbearing potential 15 Evidence of any other medical conditions (such as psychiatric illness, infectious diseases, drug or alcohol abuse, physical examination or laboratory finding) that may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment- related complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Detection (visual) of [89Zr]-Df-CriPec® docetaxel in tumour lesions (the short axis diameter of a visually assessable and quantifiable lesion must be ≥ 2 cm) | 14 days
  Visual detection (absent/present) of tumor uptake
Detection (quantitative) of [89Zr]-Df-CriPec® docetaxel in tumour lesions (the short axis diameter of a visually assessable and quantifiable lesion must be ≥ 2 cm) | 14 days
  Measured by SUVpeak values of visual positive lesions

SECONDARY OUTCOMES:
Dosimetry of [89Zr]-Df-CriPec® docetaxel | 14 days
  Based on 89Zr PK activity concentration (Bq/ml) and biodistribution [89Zr]-Df-CriPec® docetaxel scans
Optimal time point for PET imaging after [89Zr]-Df-CriPec® docetaxel administration | 14 days
  As assesed by a multidisciplinairy team
Linearity between [89Zr]-Df-CriPec® docetaxel and total docetaxel | 14 days
  Assessment of 89Zr PK (Bq/ml) and total docetaxel (ng/ml)
Biodistribution of low dose dose [89Zr]-Df-CriPec® docetaxel before and after administration of therapeutic dose of CriPec® docetaxel (quantified with %ID [89Zr] CriPec® docetaxel) | 14 days
  Measured by defining volumes of interest (VOI) of various organs on PET scan and calculating %ID/kg

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No